CLINICAL TRIAL: NCT05511727
Title: Use of Single Versus Double Foley's Catheter in Pre-induction Cervical Ripening in Postdate Primigravidae
Brief Title: Use of Single Versus Double Foley's Catheter in Pre-induction Cervical Ripening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Islam Mohamed
Record Dates: First submitted 2022-08-16; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Post Date; Induction of Labor
Keywords: primigravida; pregnants; Cervical ripening; single and double Foley's catheter
MeSH Terms: conditions — Pregnancy, Prolonged

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single Foley's catheter group (Active Comparator)
  Interventions: Device: single versus double Foley's catheter in pre-induction cervical ripening
- Double Foley's catheter group (Active Comparator)
  Interventions: Device: single versus double Foley's catheter in pre-induction cervical ripening

INTERVENTIONS:
Device: single versus double Foley's catheter in pre-induction cervical ripening — The single balloon catheter (i.e. Foley catheter [FC]) and Cook cervical ripening balloon have been the most commonly used mechanical method

SUMMARY:
Cervical ripening should be present before labor induction, which can generally be divided into two categories: pharmacological and mechanical

DETAILED DESCRIPTION:
With appropriate decision and timely intervention, labor induction decreases the risk of fetal and maternal morbidity and mortality. The single balloon catheter (i.e. Foley catheter [FC]) and Cook cervical ripening balloon have been the most commonly used mechanicalwith a minimal increase in risk of cesarean section.

The single balloon catheter (i.e. Foley catheter [FC]) and Cook cervical ripening balloon have been the most commonly used mechanical method.

The FC applies pressure on lower uterine segment and cervix in the direction from the uterus to the vagina.

The Cook cervical ripening balloon is composed of a cervicovaginal balloon and a uterine balloon. Its mechanism is similar to that of the Foley balloon, but it can apply pressure in two directions simultaneously, on both the external and internal os.

Although many studies have shown that the Cook cervical ripening balloon and FC have similar efficacy and safety.

They each have district advantages and disadvantages in labor induction. In addition to the cost advantage and wide avail- ability of the FC, the safety of labor induction with the FC has been proven by many studies.

However, some study have shown that the FC results in a higher pain score, and consequently, higher maternal request for cesarean section and higher cervical laceration incidence compared with the Cook cervical ripening balloon.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 34 years old
2. Postdate Primigravida
3. Single viable fetus.
4. Cephalic presentation.
5. Normal biophysical .
6. Bishop score of four or less.
7. RH positive women.

Exclusion Criteria:

1. Premature rupture of membranes (PROM).
2. Oligo or Polyhydramnios
3. Antepartum hemorrhage and placenta praevia.
4. Current cervical cerclage.
5. Invasive cervical carcinoma.
6. Known fetal anomaly.
7. Previous uterine scar due to myomectomy or metroplasty.
8. Cephalopelvic disproportion due to pelvic contraction or Macrosomic baby.
9. Active genital Herpes infection.
10. Chronic maternal illness.

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Cervical Ripening by using Foley's Catheter | from 0 hours to 4 hours after induction of labour
  To compare the efficacy of two mechanical devices as single and double Foley's catheter for pre-induction of labor by making cervical ripening in primigravidae whom delayed on the expected date of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine - Al-Azhar University,, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided